CLINICAL TRIAL: NCT05205512
Title: Telehealth Exercise Intervention to Improve Cardiovascular Health in Lymphoma Survivors (TECHS): A Pilot Feasibility Study
Brief Title: Telehealth Exercise Intervention to Improve Cardiovascular Health in Lymphoma Survivors, TECHS Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21595; NCI-2021-13305 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21595 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-12-27; First posted 2022-01-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (telehealth exercise) (Experimental): Patients participate in telehealth exercise intervention for 30 minutes per day, 3 days a week for 8 weeks.
  Interventions: Other: Questionnaire Administration; Other: Telemedicine
- Group II (delayed control) (Active Comparator): Patients maintain current levels of physical activity for 8 weeks. Patients may then participate in telehealth exercise intervention for 8 weeks.
  Interventions: Other: Exercise Intervention; Other: Questionnaire Administration; Other: Telemedicine

INTERVENTIONS:
Other: Exercise Intervention — Maintain current levels of physical activity
  Arms: Group II (delayed control)
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine — Participate in telehealth exercise intervention
  Other Names: Telehealth

SUMMARY:
This clinical trial tests how well a telehealth exercise intervention works to improve cardiovascular health in lymphoma survivors. Telehealth exercise is a service to help perform physical exercises at home with a care provider online. With the use of telehealth exercise lymphoma survivors may be able to participate in exercise programs safely to improve heart health and reduce the risk of cardiovascular disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of an 8-week telehealth exercise intervention, as assessed by enrollment, retention, and adherence to the telehealth exercise intervention.

SECONDARY OBJECTIVE:

I. Explore the effects of an 8-week telehealth exercise intervention on cardiovascular health, assessed by cardiopulmonary exercise test, pulmonary function test, body compositions, and blood biomarkers.

OUTLINE: Participants are randomized into 1 of 2 groups.

GROUP I (TELEHEALTH EXERCISE): Patients participate in telehealth exercise intervention for 30 minutes per day, 3 days a week for 8 weeks.

GROUP II (DELAYED CONTROL): Patients maintain current levels of physical activity for 8 weeks. Patients may then participate in telehealth exercise intervention for 8 weeks.

After completion of study treatment, participants are followed up after 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hodgkin or non-Hodgkin lymphoma.
* >= 18 years old.
* Are between 2-5 years after completing anti-cancer therapy and with no evidence of disease.
* Intermediate (4-5) to high ( >= 6) risk of cardiovascular risk factors based on six key variables: Age 30 to 50 years (y) [2]) and >= 50y [3]; anthracycline dose >250mg/m ^ 2 [1]; hypertension [2]; diabetes [2]; smoking [1]; and chest radiation [1]).
* Able to understand and sign the informed consent document.
* Physically able and willing to complete all study procedures.

Exclusion Criteria:

* Have overt cardiovascular disease within 6 months (e.g. myocardial infarction, stroke, angina).
* Have contraindications to exercise.
* Participate in structured exercise (>60 minutes/week).
* Female patients who are pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Adherence to the telehealth exercise intervention | Up to 2 years
  Adherence will be measured by the number of exercise sessions attended over the exercise sessions prescribed (17/24 sessions).

SECONDARY OUTCOMES:
Effects of an 8-week telehealth exercise intervention | At baseline up to week 9
  The physiologic effects of telehealth exercise intervention will be assessed by peak oxygen consumption (VO2) using cardiopulmonary exercise testing.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuwan Lee, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States